CLINICAL TRIAL: NCT05668936
Title: A Thorough QTc Evaluation of the Effect of Cotadutide on Cardiac Repolarization in Healthy Participants: A Randomized, Double-blind, Placebo-controlled, 3-arm Parallel Study With a Nested Crossover Design for Positive Control With Moxifloxacin Administration
Brief Title: A Thorough QTC Study to Assess the Effect of Cotadutide on Cardiac Repolarization in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinuing the development of cotadutide, a daily injectable GLP-1/glucagon co-agonist, is based on strategic pipeline considerations. The premature closure is not due to any newly observed safety signals or a change in the risk/benefit profile.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5671C00010; 2022-002479-12 (EudraCT Number)
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic fatty liver disease; Glucagon-like peptide-1 (GLP-1) receptor
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — cotadutide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Participants will receive cotadutide and will receive a single dose of moxifloxacin-placebo on Day 1 and Day 93.
  Interventions: Drug: Cotadutide; Drug: Moxifloxacin-placebo
- Arm 2A (Experimental): Participants will receive a single dose of moxifloxacin (Day 1) prior to initiating treatment with cotadutide-placebo for up to 13 weeks, followed by a single dose of moxifloxacin-placebo on Day 93.
  Interventions: Drug: Cotadutide-placebo; Drug: Moxifloxacin; Drug: Moxifloxacin-placebo
- Arm 2B (Experimental): Participants will receive a single dose of moxifloxacin-placebo (Day 1) prior to initiating treatment with cotadutide-placebo for up to 13 weeks, followed by a single dose of moxifloxacin on Day 93.
  Interventions: Drug: Cotadutide-placebo; Drug: Moxifloxacin; Drug: Moxifloxacin-placebo

INTERVENTIONS:
Drug: Cotadutide — Participants will receive a subcutaneous injection of cotadutide.
  Arms: Arm 1
Drug: Cotadutide-placebo — Participants will receive a subcutaneous injection of cotadutide-placebo.
  Arms: Arm 2A; Arm 2B
Drug: Moxifloxacin — Participants will receive a single oral dose of Moxifloxacin film-coated tablet.
  Arms: Arm 2A; Arm 2B
Drug: Moxifloxacin-placebo — Participants will receive a single oral dose of Moxifloxacin-placebo film-coated tablet.

SUMMARY:
This study will investigate the effect of multiple doses of cotadutide on the cardiac activity (QTc interval) of healthy participants.

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, placebo-controlled 3-arm parallel study with a nested crossover design for positive control with moxifloxacin administration in healthy male and female participants.

Participants will be randomized to receive treatment with either cotadutide during the 13-week treatment period (Arm 1) or cotadutide-placebo (Arm 2).

The cotadutide-placebo treatment arm will be further divided into 2 subgroups (Arms 2A and 2B), in a nested crossover design for only the placebo-treated participants.

Participants will be randomized in a 2:1:1 ratio to Arm 1, Arm 2A, and Arm 2B.

Approximately 80 participants will be randomized to have 64 evaluable participants in the study.

Each participant will be involved in the study for approximately 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants of age 18 to 55 years.
* Females must have a negative pregnancy test.
* Have a Body Mass Index (BMI) of ≥ 18 and ≤ 29.9 kg/m^2.

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition (including gastrointestinal surgery) known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of acute or chronic pancreatitis.
* Family history of sudden cardiac death before the age of 50 of a first-degree relative.
* History of additional risk factors for Torsade de Pointes (eg, heart failure, clinically important bradycardia and electrolyte disturbances eg, hypokalemia, hypocalcemia, hypomagnesemia or family history of long QT syndrome).
* History of neoplastic disease
* Any clinically significant abnormalities in clinical chemistry, hematology, urinalysis results or vital signs.
* Any clinically significant abnormalities in rhythm, conduction, or morphology of the 12-lead resting electrocardiogram (ECG).
* Any positive result on screening for serum hepatitis B surface antigen OR anti-HBc antibody, indicative of active hepatitis B (ie, participants with positive anti-HBc antibody result are acceptable if anti HBc IgM antibodies are negative), hepatitis C antibody, and Human immunodeficiency virus (HIV) antibody.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes).
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Use of drugs with enzyme-inducing properties such as St John's Wort.
* Participant has a positive test result for SARS-CoV-2 RT-PCR during screening period or at baseline.
* Participant has clinical signs and symptoms consistent with COVID-19 or a history of severe COVID-19 (hospitalization, extracorporeal membrane oxygenation, mechanically ventilated).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Time-matched change-from-baseline Fridericia's correction of QT interval (QTcF) | Up to Day 92
  Time-matched change-from-baseline QTcF after cotadutide administration compared with placebo will be assesed using a C-QTc interval analysis. The method that removes the HR dependence of the QT interval most efficiently will be chosen as the primary correction method and its corresponding change from baseline QTc will be the primary endpoint.

SECONDARY OUTCOMES:
Change from baseline in QTcF | Up to Day 94
  Change from baseline in QTcF after moxifloxacin administration compared with placebo will be assessed.
Change from baseline in Heart rate (HR) | From Day 2 up to Day 92 or early discontinuation
  The effect of cotadutide on HR will be assessed.
Change from baseline in PR interval | From Day 2 up to Day 92 or early discontinuation
  The effect of cotadutide on PR interval will be assessed.
Change from baseline in QRS interval | From Day 2 up to Day 92 or early discontinuation
  The effect of cotadutide on QRS will be assessed.
Number of participants with significant change in QTcF | From Day 2 up to Day 92 or early discontinuation
  The presence of categorical outliers for QTc after cotadutide administration will be assessed.
Number of participants with significant change in HR | From Day 2 up to Day 92 or early discontinuation
  The presence of categorical outliers for HR after cotadutide administration will be assessed.
Number of participants with significant change in PR interval | From Day 2 up to Day 92 or early discontinuation
  The presence of categorical outliers for PR after cotadutide administration will be assessed.
Number of participants with significant change in QRS interval | From Day 2 up to Day 92 or early discontinuation
  The presence of categorical outliers for QRS after cotadutide administration will be assessed.
Number of treatment-emergent changes in T-wave morphology | From Day 2 up to Day 92 or early discontinuation
  Morphological changes in the T-U complex after cotadutide administration will be investigated.
Number of treatment-emergent changes in U-waves presence | From Day 2 up to Day 92 or early discontinuation
  Morphological changes in the T-U complex after cotadutide administration will be investigated.
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) of cotadutide | Day 57 and Day 91
  AUClast as a variable of the pharmacokinetics (PK) of cotadutide will be assessed.
Area under concentration-time curve in the dose interval (AUCtau) of cotadutide | Day 57 and Day 91
  AUCtau as a variable of the PK of cotadutide will be assessed.
Maximum observed plasma concentration (Cmax) of cotadutide | Day 57 and Day 91
  Cmax as a variable of the PK of cotadutide will be assessed.
Time to reach maximum observed plasma concentration (tmax) of cotadutide | Day 57 and Day 91
  tmax as a variable of the PK of cotadutide will be assessed.
Change from baseline in mean systolic blood pressure (SBP) | Up to Day 92
  The effect of cotadutide on blood pressure (BP) by Ambulatory blood pressure monitoring (ABPM) will be investigated.
Change from baseline in mean diastolic blood pressure (DBP) | Up to Day 92
  The effect of cotadutide on BP by ABPM will be investigated.
Change from baseline in mean HR | Up to Day 92
  The effect of cotadutide on HR by ABPM will be investigated.
Placebo-corrected mean change from baseline in SBP | Up to Day 92
  The effect of cotadutide on BP by ABPM will be investigated.
Placebo-corrected mean change from baseline in DBP | Up to Day 92
  The effect of cotadutide on BP by ABPM will be investigated.
Placebo-corrected mean change from baseline in HR | Up to Day 92
  The effect of cotadutide on HR by ABPM will be investigated.
Number of participants with significant change in SBP | Up to Day 92
  The effect of cotadutide on BP by ABPM will be investigated.
Number of participants with change in DBP | Up to Day 92
  The effect of cotadutide on BP by ABPM will be investigated.
Number of participants with significant change in HR | Up to Day 92
  The effect of cotadutide on HR by ABPM will be investigated.
Number of participants with Adverse Events (AEs) | Up to follow-up visit 28 days post last dose (approximately Day 120)
  The safety and tolerability of cotadutide will be assessed.
Number of participants with Antidrug Antibodies to cotadutide | Day 2, 30, 57, 91 and Day 120 (follow-up visit 28 days post last dose)
  The immunogenicity of cotadutide will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home